CLINICAL TRIAL: NCT01162239
Title: Maintaining Nonsmoking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA002538; 2R01DA002538 (NIH); 11633 (Other: University of California, San Francisco)
Record Dates: First submitted 2010-06-14; First posted 2010-07-14 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Nicotine Dependence
Keywords: Smoking; Tobacco; Nicotine; Smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Varenicline; Medical Staff

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Extended Brief Contact (Experimental): Following standard brief treatment, participants have monthly meetings with medical staff.
  Interventions: Drug: Varenicline; Behavioral: Initial Individual counseling; Behavioral: Check-ins with medical staff
- Extended Health Education (Experimental): Following standard treatment, participants receive monthly counseling with content based on a health education model.
  Interventions: Drug: Varenicline; Behavioral: Initial Individual counseling; Behavioral: Extended Individual Counseling - Health Model
- Extended Relapse Prevention plus varenicline (Experimental): Following standard treatment, participants receive monthly counseling with content based on a relapse prevention model plus access to ongoing medication treatment with varenicline.
  Interventions: Drug: Varenicline; Behavioral: Initial Individual counseling; Behavioral: Extended Individual Counseling - Relapse Prevention Model
- Extended Relapse Prevention (Experimental): Following standard treatment, participants receive monthly counseling with content based on a relapse prevention model.
  Interventions: Drug: Varenicline; Behavioral: Initial Individual counseling; Behavioral: Extended Individual Counseling - Relapse Prevention Model

INTERVENTIONS:
Drug: Varenicline — All participants will receive 12 weeks of varenicline treatment at standard dosage of 1 mg bid. Participants in the Extended Relapse Prevention plus varenicline will receive varenicline for up to 40 additional weeks.
  Other Names: Chantix
Behavioral: Initial Individual counseling — Five 90 minute individual counseling sessions to occur during the first 12 weeks of initial treatment.
Behavioral: Check-ins with medical staff — Monthly brief (10-15 minutes) meetings with medical staff.
  Arms: Extended Brief Contact
Behavioral: Extended Individual Counseling - Health Model — Monthly counseling sessions across a nine month period with content based on a health education model. Each session is 30-45 minutes in duration.
  Arms: Extended Health Education
Behavioral: Extended Individual Counseling - Relapse Prevention Model — Eleven individual counseling sessions across a nine month period with content based on a relapse prevention model. Each session is 30-45 minutes in duration.
  Arms: Extended Relapse Prevention; Extended Relapse Prevention plus varenicline

SUMMARY:
The research is based on a chronic disorder model of cigarette smoking which suggests that long-term treatment targeted to prevent relapse may be useful. Based on this model, the investigators have developed a relapse prevention treatment to intervene on five areas important in relapse prevention, including fluctuating motivation, depression, withdrawal, weight gain, and social support. This treatment protocol has produced high long-term abstinence rates when implemented in a clinical research setting. The current study will evaluate the treatment model when implemented in a medical outpatient setting.

DETAILED DESCRIPTION:
This study will test a series of hypotheses comparing the efficacy of the relapse prevention treatment to other extended treatments. All participants will be assessed at baseline on demographics, smoking behaviors, nicotine dependence, depression, alcohol and other drug history and problems, mood disturbance, treatment support, stress, health status, and motivation for change. Participants will be randomly assigned to one of four treatment conditions. All participants will receive 12 weeks of combined pharmacological treatment (varenicline) and behavioral treatment (five individual counseling sessions). Following this brief treatment, participants will be randomly assigned to one of four treatment protocols

1. Monthly Brief Contact or
2. Extended Non-Specific Behavioral Treatment or
3. Extended Relapse Prevention Treatment or
4. Extended Relapse Prevention Treatment + availability of varenicline treatment.

Each extended treatment protocol is 40 weeks in duration following the initial 12 weeks of treatment.

All participants will be assessed at weeks 12, 24, 52, 64, and 104, on smoking as well as other psychometric measures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Must be smoking 5 or more cigarettes per day

Exclusion Criteria:

* Previous history of bipolar/manic-depressive disorder
* Current diagnosis of schizophrenia
* Acute life threatening diseases
* Evidence of alcohol or other drug abuse so severe that the patient is judged to be potentially unable to comply with the protocol
* Pregnancy or lactation
* Individuals with out of normal range blood pressure, active angina, valve disease, valve replacement, active cardiomyopathies, myocardial infarction or Coronary artery bypass grafting (CABG) within one year, and Congestive heart failure (CHF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Humfleet, Ph. D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of California, San Francisco medical clinics and the general community. Participants from the general community were recruited through flyers posted at various community health care organizations and social service agencies. Advertisements were placed in local newspapers and websites.
Pre-assignment Details: Participants were stratified based on gender, age, site, and number of cigarettes smoked per day at baseline. Participants were then randomly assigned to one of four treatment conditions derived from a double blinded allocation list prepared by a statistician. Neither participant nor the therapist were unblinded to final treatment until Week 8.
Groups:
- Extended Brief Contact: Following standard brief treatment, participants have monthly meetings with medical staff.
  Varenicline: All participants will receive 12 weeks of varenicline treatment at standard dosage of 1 mg bid.
  Individual counseling: Five 90 minute individual counseling sessions.
  Check-ins with medical staff: Monthly brief (10-15 minutes) meetings with medical staff.
- Extended Health Education: Following standard treatment, participants receive monthly counseling with content based on a health education model.
  Varenicline: All participants will receive 12 weeks of varenicline treatment at standard dosage of 1 mg bid.
  Individual counseling: Five 90 minute individual counseling sessions.
  individual counseling: Eleven individual counseling sessions across a nine month period. Each session is 30-45 minutes in duration.
- Extended Relapse Prevention Plus Varenicline: Following standard treatment, participants receive monthly counseling with content based on a relapse prevention model plus access to ongoing medication treatment with varenicline.
  Varenicline: All participants will receive 12 weeks of varenicline treatment at standard dosage of 1 mg bid.
  Individual counseling: Five 90 minute individual counseling sessions.
  individual counseling: Eleven individual counseling sessions across a nine month period. Each session is 30-45 minutes in duration.
- Extended Relapse Prevention: Following standard treatment, participants receive monthly counseling with content based on a relapse prevention model.
  Varenicline: All participants will receive 12 weeks of varenicline treatment at standard dosage of 1 mg bid.
  Individual counseling: Five 90 minute individual counseling sessions.
  individual counseling: Eleven individual counseling sessions across a nine month period. Each session is 30-45 minutes in duration.
Period: Treatment Phase
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Started | 55 | 54 | 52 | 55
Week 12 | 50 | 51 | 49 | 53
Week 24 | 51 | 48 | 48 | 50
Week 52 | 49 | 47 | 48 | 50
Completed (Treatment regimens were completed at 52 weeks) | 49 | 47 | 48 | 50
Not Completed | 6 | 7 | 4 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 5 | 4 | 2 | 1
Period: Extended Follow-up
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Started (Week 64) | 47 | 45 | 45 | 47
Completed (Week 104) | 39 | 32 | 37 | 41
Not Completed | 8 | 13 | 8 | 6
Not completed — Lost to Follow-up | 8 | 13 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention | Total
Number analyzed (Participants) | 55 | 54 | 52 | 55 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (10.8) | 53.8 (9.4) | 47.0 (11.6) | 47.3 (11.8) | 48.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 18 | 22 | 84
  Male | 34 | 31 | 34 | 33 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 1 | 8 | 26
  Not Hispanic or Latino | 43 | 44 | 49 | 46 | 182
  Unknown or Not Reported | 2 | 3 | 2 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 1 | 3 | 6 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 20 | 14 | 15 | 63
  White | 29 | 24 | 24 | 26 | 103
  More than one race | 2 | 3 | 4 | 4 | 13
  Unknown or Not Reported | 8 | 3 | 4 | 7 | 22
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 52 | 55 | 216
Number of cigarettes smoked per day [Number; unit: participants]
  10 or less cigarettes smoked per day | 14 | 10 | 14 | 15 | 55
  11 - 22 cigarettes smoked per day | 32 | 36 | 31 | 28 | 54
  21 - 30 cigarettes smoked per day | 7 | 7 | 2 | 7 | 52
  31 or more cigarettes smoked per day | 2 | 1 | 5 | 5 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at Week 12
Description: Point prevalent abstinence is defined as biochemically verified (confirmed carbon dioxide (CO) < 8 parts per million (ppm)) self-reported abstinence from smoking cigarettes in the past 7 days. Smoking status was then categorized as either Abstinent or Not Abstinent.
Time Frame: 12 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Number analyzed (Participants) | 50 | 51 | 49 | 53
Participants | 22 | 20 | 29 | 20

2. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at Week 24
Description: Point prevalent abstinence is defined as biochemically verified (confirmed carbon dioxide (CO) < 8 ppm) self-reported abstinence from smoking cigarettes in the past 7 days. Smoking status was then categorized as either Abstinent or Not Abstinent.
Time Frame: 24 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Number analyzed (Participants) | 51 | 48 | 48 | 50
Participants | 20 | 18 | 24 | 21

3. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at Week 52
Description: as for outcome 2
Time Frame: 52 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Number analyzed (Participants) | 49 | 47 | 48 | 50
Participants | 19 | 15 | 23 | 17

4. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at Follow-up Week 64
Description: as for outcome 2
Time Frame: 64 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Number analyzed (Participants) | 47 | 45 | 45 | 47
Participants | 16 | 18 | 24 | 13

5. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at Follow-up Week 104
Description: as for outcome 2
Time Frame: 104 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
Number analyzed (Participants) | 39 | 32 | 37 | 40
Participants | 16 | 13 | 16 | 13

6. Secondary Outcome: Comparison of Combined Extended vs Brief Treatment at Week 24
Description: The three extended treatment programs were combined and compared to the Brief treatment, with extended treatments expected to produce significant higher CO corrected abstinence rates overall. Comparisons will be tested using Chi-Square analysis.
Time Frame: 24 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Groups:
- Combined Extended Treatments: Patients in the extended treatments were offered the followint:
  Following standard treatment, participants receive monthly counseling with content based on a health education model.
  or
  Eleven individual counseling sessions across a nine month period plus Varenicline.Each session 30-45 minutes in duration with a focus on relapse prevention
  or
  Eleven individual counseling sessions across a nine month period. Each session 30-45 minutes in duration with a focus on relapse prevention
Arm/Group | Extended Brief Contact | Combined Extended Treatments
Number analyzed (Participants) | 51 | 146
Participants | 20 | 63
Statistical Analysis 1: Comparison: Extended Brief Contact vs Combined Extended Treatments; Test type: Other; p = 0.62, Chi-squared

7. Secondary Outcome: Comparison of Combined Extended vs Brief Treatment at Week 52
Description: as for outcome 6
Time Frame: 52 weeks following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Brief Contact | Combined Extended Treatments
Number analyzed (Participants) | 49 | 145
Participants | 19 | 55
Statistical Analysis 1: Comparison: Extended Brief Contact vs Combined Extended Treatments; Test type: Other; p = 0.91, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 104 weeks
Description: Only serious adverse events were collected for this study
Arm/Group | Extended Brief Contact | Extended Health Education | Extended Relapse Prevention Plus Varenicline | Extended Relapse Prevention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/52 | 1/55
Serious Adverse Events (participants affected / at risk) | 2/55 | 1/54 | 2/52 | 2/55
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Brief Contact (N=55) | Extended Health Education (N=54) | Extended Relapse Prevention Plus Varenicline (N=52) | Extended Relapse Prevention (N=55)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concentration Impariment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insect Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes